CLINICAL TRIAL: NCT05077267
Title: An Open Label Phase 2 Trial to Evaluate the Safety, Tolerability and Immunogenicity of the ABNCoV2 Vaccine in Severe Acute Respiratory Syndrome (SARS) Coronavirus (CoV)-2 Seronegative and Seropositive Adult Subjects
Brief Title: ABNCoV2 Vaccine in SARS-CoV-2 (COVID-19) Seronegative and Seropositive Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABNCoV2-01
Record Dates: First submitted 2021-10-11; First posted 2021-10-14 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: COVID-19 Disease
MeSH Terms: interventions — ABNCoV2 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABNCoV2 100ug single dose (Experimental): ABNCoV2 100ug single dose. Intervention type: Biological/Vaccine
  Interventions: Biological: ABNCoV2 100ug
- ABNCoV2 50ug single dose (Experimental): ABNCoV2 50ug single dose. Intervention type: Biological/Vaccine
  Interventions: Biological: ABNCoV2 50ug
- ABNCoV2 100ug two doses (Experimental): ABNCoV2 100ug two doses 4 weeks apart. Intervention type: Biological/Vaccine
  Interventions: Biological: ABNCoV2 100ug

INTERVENTIONS:
Biological: ABNCoV2 100ug — IM injection 100ug dose
  Arms: ABNCoV2 100ug single dose; ABNCoV2 100ug two doses
Biological: ABNCoV2 50ug — IM injection 50ug dose
  Arms: ABNCoV2 50ug single dose

SUMMARY:
An open label phase 2 trial to evaluate safety, tolerability and immunogenicity of the ABNCoV2 vaccine after intramuscular (IM) application. The trial will evaluate a homologous prime-boost regimen with 100 µg ABNCoV2 in initially seronegative adult subjects (Group 1), as determined by a qualitative test for SARS-CoV-2 antibodies, compared to a single boost vaccination with 100 µg (Group 2) or 50 µg (Group 3) ABNCoV2 in initially seropositive subjects, as defined by a positive qualitative test for SARS-CoV-2 antibodies and a history of SARS-CoV-2 vaccination or previous COVID-19 disease at least 90 days prior to planned trial vaccination.

DETAILED DESCRIPTION:
For this Phase 2 trial ABNCoV2-01, in a run in phase 6 adults (comprising of 3 subjects in each Group 1 and 2) will be vaccinated at 1 clinical trial site in a consecutive manner, with an at least 48 hours interval between the first and second subject of each group, then the second and third subject dosed on consecutive days, before opening up to full enrolment of the trial. Safety assessments will be based on solicited and unsolicited adverse event (AE) data (first week after vaccination) evaluated by an independent Data Monitoring Committee (DMC). After a positive DMC recommendation, enrolment to the rest of Group 1 and 2 of the trial will commence. Group 3 subjects will be enrolled after completion of Group 2 enrollment.

This phase 2 trial will evaluate a homologous prime-boost regimen with 100 µg ABNCoV2 in initially seronegative adult subjects (Group 1), as determined by a qualitative test for SARS-CoV-2 antibodies, compared to a single boost vaccination with 100 µg (Group 2) and 50 µg (Group 3) ABNCoV2 in initially seropositive subjects, as defined by a positive qualitative test for SARS-CoV-2 antibodies and either a history of SARS-CoV-2 vaccination or previous COVID-19 disease (Group 2 and 3) at least 90 days prior to planned trial vaccination.

Due to the timing of the addition of Group 3, enrollment into Group 2 will be completed prior to enrolling subjects into Group 3. Therefore, no randomization will be required for the seropositive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Seronegative (Group 1): negative qualitative test for SARS-CoV-2 antibodies at SCR.

Seropositive (Group 2 and Group 3): Previous COVID-19 disease or previously completed vaccination regimen with an authorized SARS-CoV-2 vaccine at least 90 days before planned trial vaccination and a positive qualitative test for SARS-CoV-2 antibodies at SCR. "Authorized" SARS-CoV-2 vaccine refers to authorization status at SCR, i.e., subjects can be eligible if the subject previously received investigational vaccines that have since been authorized for emergency use or granted full market licensure. Receipt of a single dose of an authorized COVID-19 vaccine regimen in subjects with a previous diagnosis of COVID-19 or a mix/match series of 2 doses of any authorized COVID-19 vaccine will be considered as a completed vaccination.

* General good health, without acute medical illness, physical exam findings, or laboratory abnormalities, as determined by the investigator.
* Body mass index (BMI) ≥18.5 and <40.
* Female subjects of childbearing potential (WOCBP) must agree to the use of an effective method of birth control from at least 30 days prior to administration of the vaccine until 30 days after the vaccination. Male subjects who are sexually active with a WOCBP must agree to the use of an effective method of birth control from the day of administration of the vaccine until 30 days after the vaccination.
* Negative human immunodeficiency virus antibody test (anti HIV), negative hepatitis B surface antigen (HBsAG) and negative antibody to hepatitis C virus (HCV).

Exclusion Criteria:

• Group 1 only: History of COVID-19 infection or previous vaccination with a licensed or candidate SARS-CoV-2 vaccine, or positive qualitative test for SARS-CoV-2 antibodies at SCR.

Groups 2 and 3 only: History of COVID-19 infection and subsequent receipt of more than one licensed or candidate SARS-CoV-2 vaccine.

* Positive test for SARS-CoV-2 infection at SCR.
* Pregnant or breastfeeding women.
* Subject has an acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of the responses.
* History of or active autoimmune disease. History of Guillain-Barré syndrome or Reye's syndrome. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
* Known or suspected impairment of immunologic functions including, but not limited to, known immunodeficiency syndrome.
* History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months prior to SCR that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous tumor site.
* Laboratory parameters (such as complete blood count, serum biochemistry including aspartate aminotransferase (AST), alanine amino transferase (ALT), alkaline phosphokinase (AP), bilirubin, or creatinine values), pulse rate, blood pressure, or electrocardiogram (ECG) outside normal range at SCR and deemed clinically relevant by the investigator.
* Clinically significant mental disorder not adequately controlled by medical treatment.
* Active or recent history (within 6 months before SCR) of chronic alcohol abuse, intravenous drug abuse, or nasal drug abuse.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis or severe allergic reaction to any vaccine.
* Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after trial vaccination.
* Having received any vaccinations or planned vaccinations with an inactivated vaccine within 14 days prior to or after trial vaccination.
* Recent blood donation (including platelets, plasma and red blood cells) within 4 weeks prior to SCR, or planned blood donations during the active trial phase.
* Chronic systemic administration (defined as more than 14 days of >5 mg prednisone [or equivalent]/day), or any other immune-modifying drugs during a period starting 3 months prior to administration of the vaccine and ending 4 weeks after the last vaccination. The use of topical, inhaled, ophthalmic and nasal glucocorticoids is allowed.
* Post organ transplant subjects, whether or not receiving chronic immunosuppressive therapy.
* Administration or planned administration of immunoglobulins and/or any blood products during a period starting 3 months prior to administration of the vaccine and ending 4 weeks after the last vaccination. Receipt of packed red blood cells given for an emergency indication in an otherwise healthy person, and not required as ongoing treatment is not exclusionary (for example packed red blood cells given in emergency during an elective surgery).
* Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the administration of trial vaccine, or planned administration of such a drug or vaccine throughout the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Grigat, MD, Principal Investigator — Velocity Clinical Research Hamburg
Locations (2):
- Germany (2):
  - Emovis GmbH, Berlin
  - Velocity Clinical Research Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 210 subjects were to be enrolled in this trial, beginning with a run-in phase of 6 subjects (3 in each of Groups 1 and 2) before enrollment opened to both treatment groups pending positive results from a safety Data Monitoring Committee. Enrollment was based on prior SARS-CoV-2 experience, with Group 1 being seronegative and Group 2 being seropositive. Group 3 was enrolled after completion of the prior groups with a lower dose level for seropositive subjects.
Groups:
- Group 1: Seronegative adult subjects 100ug ABNCoV2 by subcutaneous injection on Day 1 and Day 29
- Group 2: Seropositive adult subjects 100ug ABNCoV2 by subcutaneous injection on Day 1
- Group 3: Seropositive adult subjects 50ug ABNCoV2 by subcutaneous injection on Day 1
Period: Treatment Period
Arm/Group | Group 1 | Group 2 | Group 3
Started | 28 | 103 | 66
Completed | 28 | 101 | 66
Not Completed | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Follow-up Period
Arm/Group | Group 1 | Group 2 | Group 3
Started (Subject could participate in follow-up even if not completing the treatment period.) | 28 | 103 | 66
Completed | 28 | 3 | 0
Not Completed | 0 | 100 | 66
Not completed — Lost to Follow-up | 0 | 5 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 5
Not completed — Study terminated by sponsor | 0 | 27 | 23
Not completed — Received COVID-19 booster outside of trial | 0 | 66 | 30
Not completed — Patient is busy at work and withdraws the IC | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one vaccination with ABNCoV2 at any time during the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 28 | 103 | 66 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 79 | 59 | 165
  >=65 years | 1 | 24 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (12.72) | 51 (15.88) | 46.3 (14.39) | 48.7 (15.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 42 | 33 | 92
  Male | 11 | 61 | 33 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 28 | 103 | 65 | 196
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 24 | 100 | 65 | 189
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Germany | 28 | 103 | 66 | 197

OUTCOME MEASURES:

1. Primary Outcome: Severe Acute Respiratory Syndrome (SARS) Coronavirus (CoV)-2 Index Virus Neutralizing Antibody Titers at 2 Weeks After the Last Vaccination
Description: The primary endpoint was SARS-CoV-2 index virus neutralizing antibody titers by pseudovirus assay at 2 weeks after the last vaccination, i.e., after the second vaccination in initially seronegative subjects (Group 1) and after the single boost vaccination in initially seropositive subjects (Groups 2 and 3), for subjects in the Immunogenicity Analysis Set.
Time Frame: 2 weeks after the second vaccination in initially seronegative subjects (Group 1) and after the single boost vaccination in initially seropositive subjects (Groups 2 and 3)
Population: All subjects who were in the Safety Analysis Set and had at least 1 post-vaccination neutralizing antibody titer result. Subjects with protocol deviations substantially affecting the immunogenicity outcomes were excluded from this analysis set. For the purpose of the primary estimate, this included SARS-CoV-2 infection prior to 2 weeks after last vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 24 | 99 | 65
titer | 516.7 [309.0 to 864.0] | 970.9 [804.1 to 1172.3] | 978.9 [781.0 to 1226.8]

2. Secondary Outcome: Subjects Reporting Any SAEs or AESIs Assessed as Related to Trial Vaccine Within 8 Days After Vaccination
Description: Subjects reporting any serious adverse events (SAEs) or adverse events of special interest (AESIs) assessed as related to trial vaccine within 8 days after vaccination
Time Frame: Within 8 days of the Day 1 vaccination for Groups 1, 2, and 3, as well as within 8 days of the Day 29 vaccination for Group 1.
Population: All subjects who received at least one vaccination with ABNCoV2 at any time during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 28 | 103 | 66
Participants | 0 | 0 | 0

3. Secondary Outcome: Subjects Reporting Any Grade ≥ 3 AEs Assessed as Related to Trial Vaccine Within 8 Days After Vaccination
Description: Subjects reporting any Grade ≥ 3 adverse events (AEs) assessed as related to trial vaccine within 8 days after vaccination
Time Frame: as for outcome 2
Population: All subjects who received at least one vaccination with ABNCoV2 at any time during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 28 | 103 | 66
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Overall trial from first vaccination through final follow up visit; i.e., 17 weeks for Group 1 and 2 years for Groups 2 and 3.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/103 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/28 | 5/103 | 1/66
Other Adverse Events (participants affected / at risk) | 9/28 | 7/103 | 3/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=28) | Group 2 (N=103) | Group 3 (N=66)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=28) | Group 2 (N=103) | Group 3 (N=66)
Nasopharyngitis (Infections and infestations) | 5 (6) | 7 (7) | 3 (3)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator agree to submit any proposed publication or presentation to Sponsor for review at least 60 days prior to submitting any such proposed publication to a publisher or proceeding with such proposed presentation. Sponsor shall have the right to require Institution/Investigator to remove specifically identified Confidential Information and/or to delay the proposed publication or presentation for an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (2):
  • Study Protocol (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT05077267/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT05077267/SAP_001.pdf